CLINICAL TRIAL: NCT02298608
Title: The Efficacy and Safety of Irreversible Electroporation for the Ablation of Renal Masses: A Prospective, Human, In-Vivo Study.
Brief Title: Efficacy and Safety of IRE for RMs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, P.G.K. Wagstaff, M.D., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL 44785.018.13
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Kidney Cancer
Keywords: Renal mass; Kidney cancer; Irreversibel Electroporation; Ablation; Safety; Efficacy; IRE
MeSH Terms: conditions — Kidney Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irreversible Electroporation (Experimental): Percutaneous, CT guided, Irreversible Electroporation of renal mass
  Interventions: Device: Nano Knife

INTERVENTIONS:
Device: Nano Knife — Percutaneous, CT guided, ablation of renal mass
  Other Names: Irreversible Electroporation

SUMMARY:
Background:

Electroporation or electropermeabilisation is a novel technique with the potential to overcome the main disadvantages of thermal ablation. It utilizes electric pulses, traveling between two or more electrodes, to create 'nanopores' in the cell membrane. If the applied current reaches a certain threshold these 'nanopores' become permanent resulting in cell death. The use of electric current means that IRE is not susceptible to 'thermal sink' leading to consistent ablation results. IRE ablation targets the cell membrane, sparing tissue architecture and minimizing damage to blood vessels, nerves and the renal collecting system.

The first in human studies have proven the safety of IRE for the ablation of small renal masses. However the efficacy of IRE through histopathological examination of an ablated renal tumour has not yet been studied, compromising the correct and scientific evaluation of this new technology.

Primary Objectives:

* To determine the efficacy of IRE ablation of renal masses , measured by histopathologic examination of the targeted tumour.
* To determine the safety of IRE ablation of renal masses, by evaluating device and procedural adverse events.

Secondary Objectives:

* To evaluate the efficacy of MRI in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation.
* To evaluate the efficacy of CEUS in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation.

Population:

10 patients, age ≥ 18 years, presenting with a solid enhancing mass, who are candidates for radical nephrectomy.

Intervention:

Eligible patients will receive IRE ablation of their renal mass 4 weeks prior to radical nephrectomy. Follow-up at one and four weeks post IRE will be performed using MRI and CEUS imaging. After radical nephrectomy histopathological examination will be performed to evaluate IRE ablation success.

DETAILED DESCRIPTION:
Rationale:

The past decades have shown an increase in the incidence of small renal masses (SRM). At the moment laparoscopic partial nephrectomy is the 'golden standard' in treatment of SRMs. Thermal ablation techniques are indicated in patients who are poor surgical candidates or who have a predisposition to develop multiple tumours. Recent studies have shown thermal ablation techniques to have similar long-term oncologic results. Downsides to thermal ablation are the possible damage to vital structures in the vicinity of the ablation zone, e.g. collecting system or intestine, and unpredictable results due to difficulty in monitoring the ablation zone and 'thermal sink'.

Electroporation or electropermeabilisation is a novel technique with the potential to overcome the main disadvantages of thermal ablation. It utilizes electric pulses, traveling between two or more electrodes, to create 'nanopores' in the cell membrane. If the applied current reaches a certain threshold these 'nanopores' become permanent resulting in cell death. The use of electric current means that IRE is not susceptible to 'thermal sink' leading to consistent ablation results. IRE ablation targets the cell membrane, sparing tissue architecture and minimizing damage to blood vessels, nerves and the renal collecting system.

The first in human studies have proven the safety of IRE for the ablation of small renal masses. However the efficacy of IRE through histopathological examination of an ablated renal tumour has not yet been studied, compromising the correct and scientific evaluation of a new technology. This is the primary objective of this research project.

Objectives:

Primary Objectives:

* To determine the efficacy of IRE ablation of renal masses , measured by histopathologic examination of the targeted tumour.
* To determine the safety of IRE ablation of renal masses, by evaluating device and procedural adverse events.

Secondary Objectives:

* To evaluate the efficacy of MRI in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation.
* To evaluate the efficacy of CEUS in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation.

Study design:

This is a prospective, human, in-vivo pilot study. Study population: 10 patients, age ≥ 18 years, presented with a solid enhancing RM , who are candidates for radical nephrectomy.

Intervention:

Patients will receive IRE ablation of the RM, performed under general anaesthesia, 4 weeks before radical nephrectomy. Follow-up at one and four weeks post IRE will be performed using MRI and CEUS imaging. After radical nephrectomy histopathological examination will be performed to evaluate IRE ablation success.

Main study parameters/endpoints:

Primary endpoints:

* The efficacy of IRE ablation of renal masses , measured by histopathologic examination of the targeted tumour by an experienced genitourinary pathologist. Using immunehistochemical staining to evaluate cell viability.
* The safety of IRE ablation of renal masses, by evaluating device and procedural adverse events using CTCAE v4.0.

Secondary endpoints:

* The efficacy of MRI in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation. By comparing MRI imaging to the histopathological examination results of the resected material.
* The efficacy of CEUS in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation. By comparing CEUS imaging to the histopathological examination results of the resected material.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

There are no benefits for patients that participate in this study. Study participants will be exposed to additional risk when compared to standard treatment. They will have to undergo an additional procedure under general anaesthesia with muscle relaxation. The exposure to ionizing radiation during the procedure has been estimated at 32 mSv. Patients have to be informed about the risks of procedural complications. Information on the efficacy of IRE, proven histopathologically, is a vital step in order to progress to long term follow-up studies without tumour excision. So far no study has investigated the efficacy of IRE for the ablation of renal tumours in this manner.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Solid, enhancing mass on cross sectional imaging
* Scheduled for a radical nephrectomy, open or laparoscopic.
* Signed informed consent

Exclusion Criteria:

* Irreversible bleeding disorders
* Inability/unwillingness to interrupt anticoagulation therapy
* Previous cryoablation, RFA or partial nephrectomy in affected kidney
* Anaesthesia Surgical Assignment (ASA), category ≤ IV
* ICD / pacemaker
* Severe cardiovascular disease in medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of IRE ablation of renal masses , measured by histopathologic examination of the targeted tumour by an experienced genitourinary pathologist. Using immunehistochemical staining to evaluate cell viability. | 1 month
Number of device and procedural adverse events using CTCAE v4.0. | 1 month

SECONDARY OUTCOMES:
The efficacy of MRI in the imaging of ablation success | 1 month
  The efficacy of MRI in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation. By comparing MRI imaging to the histopathological examination results of the resected material.
The efficacy of CEUS in the imaging of ablation success | 1 month
  The efficacy of CEUS in the imaging of ablation success, extend of the ablation zone, one and four weeks post IRE ablation. By comparing CEUS imaging to the histopathological examination results of the resected material.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. M. Pilar Laguna Pes, M.D. Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Prof. Jean J de la Rosette, M.D. Ph.D., Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Dept. Urology, Academic Medical Center, Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Wagstaff PG, de Bruin DM, Zondervan PJ, Savci Heijink CD, Engelbrecht MR, van Delden OM, van Leeuwen TG, Wijkstra H, de la Rosette JJ, Laguna Pes MP. The efficacy and safety of irreversible electroporation for the ablation of renal masses: a prospective, human, in-vivo study protocol. BMC Cancer. 2015 Mar 22;15:165. doi: 10.1186/s12885-015-1189-x. PMID 25886058